CLINICAL TRIAL: NCT04425421
Title: Recommendations for the Treatment of Children With Burkitt's Lymphoma
Acronym: GFALMB2019
Status: Recruiting | Type: Observational
Sponsor: French Africa Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: GFA LMB 2019
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Burkitt Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: OBSERVATIONAL — OBSERVAITON OF THE CAPACITY OF THE GROUP TO TREAT ACCORDING TO THE PROTOCOLE AND LOOK AT OUTCOME FOR STAGE I AND II DISEASE

SUMMARY:
This is the 4th LMB study by the French African Pediatric Oncology Group (GFAOP). The study hopes to be able to evaluate children earlier with stage I and II disease and to evaluate treatment response earlier so that the units can decide if a change in treatment is necessary, it is also hoped to provide an intensification of treatment for the stage IV disease.

DETAILED DESCRIPTION:
This is the 4th Burkitt's Lymphoma (LMB) study by the GFAOP group. This study hopes to include at least 14 Sub Saharian countries some of whom have never participated in a LMB study. The evaluation of improvement in early diagnosis should be possible in this study. The study hopes to be able to evaluate children earlier, with stage I and II disease and to evaluate treatment response earlier so that the units can decide if a change in treatment is necessary, it is also hoped to provide an intensification of treatment for children with a stage IV disease.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Burkitt's Lymphoma: all location. Diagnosis by cytology or histology. Not possible to follow all the treatment.

-

Exclusion Criteria:

Not a B Cell tumor. Child has been previously treated. Child has also another illness which would render the treatment incompatible. Parents refusal.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All Children with a Burkitt's Lymhoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the number of cases with local disease. | 5 years
  evaluating the initial clinical reports and later histological reports to confirm the diagnosis and the stage.
Evaluation of the number of cases by stage at the time of diagnosis. | 5 Years
  evaluating the initial clinical reports and later histological reports to confirm the stage and the diagnosis.
Evaluating the treatment given. | 5 Years
  Comparison of treatment given and recommended treatment.
Evaluating the follow up after treatment. | 5 Years
  How many children alive or dead after treatment
Number of relapse cases | 5 years
  The evaluation and the treatment of relapse and outcome

SECONDARY OUTCOMES:
Application of therapeutic recommendations | 5 years
  Evaluations of the correct application of recommendations

CONTACTS AND LOCATIONS:
Locations (7):
- Hopital Yalgado Ouedraogo, Ouagadougou, Burkina Faso
- CHU de Treichville à ABIDJAN, Abidjan, Côte d’Ivoire
- Democratic Republic of the Congo (2):
  - Cliniques Universitaires de Kinshasa, Kinshasa, Kinshasa City
  - Cliniques Universitaires de Lubumbashi (CUL), Lubumbashi
- HJRA, Hôpital universitaire Joseph Ravoahangy Andrianavalona, Antananarivo, Madagascar
- CHU Gabriel Touré (HGT), Bamako, Mali
- Hôpital Aristide Le Dantec, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided